CLINICAL TRIAL: NCT02260297
Title: A Study of Wrist Actigraphy in Overweight and Obese Adults With Sleep Disorders
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Guang Ning, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CCEMD-023
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Sleep Disorders
Keywords: Actigraphy; overweight and obese adults; sleep disorders
MeSH Terms: conditions — Sleep Wake Disorders; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Wrist Actigraphy(motion sensors)with light sensors-Jawbone Up 2

SUMMARY:
70 overweight or obese adults with sleep disorders will be recruited for this study, in which the investigators aim to compare wrist actigraphy with polysomnography (PSG) for sleep monitoring. It is to evaluate the applications of Jawbone Up2 with the sleep parameters derived from this actigraphy.

DETAILED DESCRIPTION:
As an observation study, it will recruit 70 overweight or obese patients with sleep disorders who meet the selection criteria: clinical records and AIS at a tertiary hospital. The patients will sign the informed consent form. The involved patients and doctors will receive related training.

These patients will receive the sleep monitoring from 21:00 to 6:00 in sleep monitoring laboratory in Ruijin Hospital. They will receive the PSG and Jawbone Up 2 sleep monitoring at the same time. Sleep parameters derived from actigraphy and PSG will be compared in multiple night recordings such as total sleep time, wake after sleep onset, sleep onset latency, awakening, sleep efficiency, total time in bed,. The aim is to assess the validation of actigraphy in overweight or obese patients with sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have one or more sleep disorders such as consecutive snoring, insomnia, sleep apnea, narcolepsy, delayed sleep phase syndrome
* Athens Insomnia Scale (AIS)>6
* BMI>25
* Agree to participate in the study and have signed the inform consent form

Exclusion Criteria:

* Terminal illness
* Physically-challenged and paralyzed patients
* Intend to receive selective surgery, to get pregnancy and breast feeding in three months
* Long-term use of the sleeping pills
* Hearing loss or severe visual disorder;
* Mental disorders
* Dementia or communication disorders
* Unable to complete an all night sleep monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight and obese adults with sleep disorders
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time, TST | 10 hrs
Wake After Sleep Onset, WASO | 10 hrs

SECONDARY OUTCOMES:
Sleep Onset Latency, SOL | 10 hrs
Frequency of arousal during sleep,awakenings | 10 hrs
Sleep Efficiency, SE | 10 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China